CLINICAL TRIAL: NCT05014815
Title: AdvanTIG-205: A Phase 2, Randomized Study of Ociperlimab (BGB-A1217) and Tislelizumab With Chemotherapy in Patients With Previously Untreated Locally Advanced, Unresectable, or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Ociperlimab With Tislelizumab and Chemotherapy in Participants With Untreated Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AdvanTIG-205; 2021-001075-17 (EudraCT Number); CTR20212782 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced, Unresectable, or Metastatic Nonsmall Cell Lung Cancer (NSCLC); Nonsmall Cell Lung Cancer, Stage IIIB; Nonsmall Cell Lung Cancer, Stage IV
Keywords: metastatic; Lung Cancer; Non-Squamous; Ociperlimab; Tislelizumab; Anti-PD-1; BGB-A317; BGB-A1217; Anti-TIGIT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Lung Neoplasms | interventions — tislelizumab; Carboplatin; Paclitaxel; Taxes; Cisplatin; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (O+T+C) (Experimental): During the induction phase, participants received ociperlimab (O) 900 mg IV, tislelizumab (T) 200 mg IV, and histology-based chemotherapy (C) every 21 days for 4-6 cycles. For squamous NSCLC, chemotherapy included carboplatin AUC 5 or 6 (on Day 1) + paclitaxel 175 or 200 mg/m² (Day 1) or nab-paclitaxel 100 mg/m² (Days 1, 8, 15) every 3 weeks. For non-squamous NSCLC, chemotherapy included cisplatin 75 mg/m² or carboplatin AUC 5 (Day 1) + pemetrexed (P) 500 mg/m² IV (Day 1), every 3 weeks.
  In the maintenance phase, non-squamous NSCLC participants received O 900 mg IV, T 200 mg IV, and pemetrexed 500 mg/m² IV every 3 weeks. Squamous NSCLC participants received O 900 mg IV and T 200 mg IV every 3 weeks until toxicity, consent withdrawal, or investigator-determined lack of benefit.
  Interventions: Drug: Ociperlimab; Drug: Tislelizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Cisplatin; Drug: Pemetrexed
- Arm B (P+T+C) (Placebo Comparator): During the induction phase, participants received placebo (P) 900 mg IV, tislelizumab (T) 200 mg IV, and histology-based chemotherapy (C) every 21 days for 4-6 cycles. For squamous NSCLC, chemotherapy included carboplatin AUC 5 or 6 (Day 1) + paclitaxel 175 or 200 mg/m² (Day 1) or nab-paclitaxel 100 mg/m² (Days 1, 8, 15) every 3 weeks. For non-squamous NSCLC, chemotherapy included cisplatin 75 mg/m² or carboplatin AUC 5 (Day 1) + pemetrexed (P) 500 mg/m² IV (Day 1), every 3 weeks.
  In the maintenance phase, non-squamous NSCLC participants received placebo 900 mg IV, T 200 mg IV, and pemetrexed 500 mg/m² IV every 3 weeks. Squamous NSCLC participants received placebo IV and T 200 mg IV every 3 weeks until toxicity, consent withdrawal, or investigator-determined lack of benefit.
  Interventions: Drug: Tislelizumab; Drug: Carboplatin; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: Cisplatin; Drug: Pemetrexed; Drug: Placebo

INTERVENTIONS:
Drug: Ociperlimab — 900 mg intravenously (IV) once every 3 weeks (Q3W)
  Other Names: BGB-A1217
  Arms: Arm A (O+T+C)
Drug: Tislelizumab — 200 mg IV Q3W
  Other Names: BGB-A317
Drug: Carboplatin — Area under the concentration-time curve (AUC) of 5 or 6, administered on Day 1 of each 21-day cycle
Drug: Paclitaxel — 75 or 200 mg per square meter (mg/m²) of body surface area, administered on Day 1 of each 21-day cycle
Drug: Nab paclitaxel — 100 mg/m², administered intravenously on Days 1, 8, and 15 of each 21-day cycle
Drug: Cisplatin — 75 mg/m², administered intravenously on Day 1 of each 21-day cycle
Drug: Pemetrexed — 500 mg/m² administered intravenously on Day 1 of each 21-day cycle
Drug: Placebo — Administered intravenously Q3W to match ociperlimab
  Arms: Arm B (P+T+C)

SUMMARY:
This study aimed to evaluate the safety and effectiveness of ociperlimab combined with tislelizumab and chemotherapy, compared to tislelizumab and chemotherapy alone, in participants with non-small cell lung cancer (NSCLC) that was locally advanced, could not be removed by surgery, or had spread to other parts of the body.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants had histologically or cytologically confirmed locally advanced or recurrent non-small cell lung cancer (NSCLC) that was not eligible for curative surgical resection and/or definitive radiotherapy, with or without chemotherapy. Alternatively, participants had metastatic non-squamous or squamous NSCLC.
2. Participants had not received any prior systemic therapy for locally advanced or metastatic squamous or non-squamous NSCLC, including but not limited to chemotherapy or targeted therapies. Those who had previously received neoadjuvant or adjuvant chemotherapy, or chemoradiotherapy with curative intent for non-metastatic disease, were required to have experienced a disease-free interval of at least 6 months from the last dose of chemotherapy and/or concurrent radiotherapy prior to randomization.
3. Archival tumor tissue or a fresh biopsy (if archival tissue was unavailable) was required for programmed death-ligand 1 (PD-L1) level assessment and retrospective biomarker analyses. Only participants with evaluable PD-L1 results were considered eligible.
4. Participants were required to have had at least one measurable lesion as assessed by the investigator in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Participants had an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

Key Exclusion Criteria:

1. Participants were excluded if they had known mutations in any of the following genes:

   * Epidermal Growth Factor Receptor (EGFR): For participants with non-squamous NSCLC and unknown EGFR mutation status, tissue-based EGFR testing (performed either locally or at a central laboratory) or an endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA)-based EGFR test was required prior to enrollment. Those found to harbor EGFR-sensitizing mutations were excluded.
   * Anaplastic Lymphoma Kinase (ALK) fusion oncogene.
   * B-Raf Proto-Oncogene (BRAF) V600E mutation.
   * ROS Proto-Oncogene 1 (ROS1) rearrangement.
2. Participants who had received prior treatment with EGFR inhibitors, ALK inhibitors, or other targeted therapies for known driver mutations.
3. Participants who had received any prior therapies targeting T-cell costimulatory or checkpoint pathways (e.g., programmed cell death protein 1 [PD-1], programmed death-ligand 1 [PD-L1], or cytotoxic T-lymphocyte-associated protein 4 [CTLA-4]) for metastatic NSCLC were excluded.
4. Participants who had any condition requiring systemic treatment with corticosteroids at a dose greater than 10 mg of prednisone (or equivalent) daily, or other immunosuppressive medications within 14 days prior to randomization.
5. Participants who had an active infection, including but not limited to tuberculosis, requiring systemic antibacterial, antifungal, or antiviral treatment within 14 days prior to randomization were excluded.

Note: Additional protocol-defined inclusion and exclusion criteria may have applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (64):
- United States (11):
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Rj Zuckerberg Cancer Center, New Hyde Park, New York
  - North Shore Hematology Oncology Associates Dba New York Cancer and Blood Specialists (New York), New York, New York
  - North Shore Hematology Oncology Associates Dba New York Cancer and Blood Specialists, Port Jefferson Station, New York
  - Ny Cancer and Blood Specialists, The Bronx, New York
  - Xcancerdayton Physician Network, Dayton, Ohio
  - Tennessee Cancer Specialist, Knoxville, Tennessee
  - Texas Oncology Tyler Longview, Austin, Texas
  - Cancer Care Northwest, Spokane Valley, Washington
- Australia (8):
  - Border Medical Oncology, East Albury, New South Wales
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Townsville University Hospital, Douglas, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Launceston General Hospital, Launceston, Tasmania
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Olivia Newton John Cancer Wellness and Research Centre, Heidelberg, Victoria
- Klinik Penzing Wien, Abteilung Fur Atemwegs, Vienna, Austria
- China (24):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital Affiliated to the Army Medical University, Chongqing, Chongqing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - The First Peoples Hospital of Chenzhou, Chenzhou, Hunan
  - Changzhou Cancer Hospital, Changzhou, Jiangsu
  - Ansteel Group General Hospital, Anshan, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Liaocheng Peoples Hospital, Liaocheng, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The First Peoples Hospital of Kashgar, Kashgar, Xinjiang
  - Zhejiang Provincial Peoples Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
- France (4):
  - Centre Hospitalier Regional Universitaire de Caen, Caen
  - Institut Curie, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Charles Nicolle Clinique Pneumologique, Rouen
- St Lukes Hospital, Thessaloniki, Greece
- South Korea (10):
  - Dong A University Hospital, Seogu, Busan Gwang'yeogsi
  - Cha Bundang Medical Center, Cha University, BundangGu SeongnamSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Korea University Guro Hospital, GuroGu, Seoul Teugbyeolsi
  - Kangbuk Samsung Hospital, JongnoGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Ulsan University Hospital, Donggu, Ulsan Gwang'yeogsi
  - Ajou University Hospital, Suwon
- Spain (5):
  - Centro Oncologico de Galicia, A Coruña
  - Ch Provincial de Castellon, Castellon
  - Complejo Asistencial Universitario de Leon, León
  - Hospital Universitario Central de Asturias, Oviedo
  - Fundacion Instituto Valenciano de Oncologia Ivo, Valencia

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved. BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations. Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 75 study centers in 8 countries (China, South Korea, United States of America, Australia, France, Spain, Austria, Greece).
Pre-assignment Details: Eligible participants were randomized in a 1:1 ratio to receive either ociperlimab or placebo treatment, plus tislelizumab and chemotherapy. Randomization was stratified by histology (squamous versus non--squamous), and programmed cell death protein ligand-1 (PD-L1) expression.
Groups:
- Arm A (O+T+C): Ociperlimab (900 mg IV), tislelizumab (200 mg IV), and histology-based chemotherapy
- Arm B (P+T+C): Placebo, tislelizumab (200 mg IV), and histology-based chemotherapy
Period: Overall Study
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
Started | 136 | 136
Treated | 135 | 136
Completed | 57 | 50
Not Completed | 79 | 86
Not completed — Death | 63 | 70
Not completed — Withdrawal by Subject | 10 | 10
Not completed — Lost to Follow-up | 4 | 2
Not completed — Physician Decision | 2 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat Analysis Set is defined as all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C) | Total
Number analyzed (Participants) | 136 | 136 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.02 (8.006) | 63.77 (9.366) | 63.90 (8.697)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 32 | 54
  Male | 114 | 104 | 218
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 105 | 102 | 207
  Black or African American | 0 | 1 | 1
  White | 23 | 25 | 48
  Not Reported | 8 | 7 | 15
  Unknown | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 123 | 123 | 246
  Hispanic or Latino | 1 | 4 | 5
  Not Reported | 8 | 7 | 15
  Unknown | 4 | 2 | 6
Histology [Count of Participants; unit: Participants] — Histology stratification refers to the classification of participants based on tumor cell morphology. Squamous histology is defined by malignant transformation of flat epithelial cells typically lining the airways, while nonsquamous histology includes adenocarcinoma, large cell carcinoma, and other subtypes arising from glandular or poorly differentiated epithelial cells.
  Participants
    Squamous | 55 | 56 | 111
    Non-Squamous | 81 | 80 | 161
Programmed Death-Ligand 1 (PD-L1) Expressio [Count of Participants; unit: Participants] — PD-L1 is a protein that can help cancer cells avoid being killed by the immune system. PD-L1 score was based on the % of tumor area with PD-L1-stained tumor or immune cells, using the TAP (Tumor Area Positive) Score method, previously called vCPS. Scores were obtained via Interactive Response Technology.
  Participants
    < 1% of tumor cells | 57 | 58 | 115
    1-49% of Tumor Cells | 42 | 42 | 84
    > 50% of Tumor Cells | 37 | 36 | 73

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the first objectively documented disease progression as assessed by the investigator per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v1.1) or death from any cause, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 04 September 2024; Up to 33 months
Population: Intent-To-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
Number analyzed (Participants) | 136 | 136
Months | 8.2 [6.2 to 10.6] | 8.1 [6.0 to 10.2]
Statistical Analysis 1: Comparison: Arm A (O+T+C) vs Arm B (P+T+C); Test type: Superiority; p = 0.4698, Log Rank — 1-sided p-value; Stratified by PD-L1 expression (<1% of tumor cells (TC) vs 1-49% TC vs >= 50% TC) and histology (squamous vs non-squamous); Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.74 to 1.33] — The HR and its 95% confidence interval (CI) was estimated using a Cox regression model stratified by PD-L1 expression (<1% of tumor cells (TC) vs 1-49% TC vs >= 50% TC) and histology (squamous vs non-squamous)

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the percentage of participants who had a confirmed complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 Tumor assessments.
  CR is defined as the disappearance of all target and non-target lesions and no new lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 04 September 2024; Up to 33 months
Population: Intent-To-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
Number analyzed (Participants) | 136 | 136
percentage of participants | 41.9 [33.5 to 50.7] | 47.8 [39.2 to 56.5]
Statistical Analysis 1: Comparison: Arm A (O+T+C) vs Arm B (P+T+C); Test type: Other; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.47 to 1.26] — The Mantel-Haenszel common OR and its 95% CI were estimated using a normal approximation of the log odds ratio and the Robins-Breslow-Greenland variance, stratified by PD-L1 expression and histology

3. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first documented objective response to documented radiological disease progression as assessed by the investigator using RECIST v1.1, or death from any cause, whichever occurred first. Median DOR was estimated using the Kaplan-Meier method.
  Progressive disease is captured as at least a 20% increase in the sum of diameters of target lesions, using the smallest sum on study as the reference (including the baseline sum if it was the smallest). In addition to the 20% relative increase, the sum also had to show an absolute increase of at least 5 mm.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 04 September 2024; Up to 33 months
Population: The analysis included only intent-to-treat participants with a confirmed complete or partial response per RECIST v1.1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
Number analyzed (Participants) | 57 | 65
months | 10.4 [8.0 to 17.7] | 11.2 [8.1 to 13.9]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the documented date of death for participants who died on or before the clinical cutoff date. Median OS was calculated using the Kaplan-Meier method. Data for participants who were alive at the clinical cutoff date were censored at their last known alive date, defined as either the clinical cutoff date for those still on treatment or the most recent available date confirming they were alive, whichever occurred first.
Time Frame: From randomization up to the final efficacy analysis data cut-off date of 04 September 2024; Up to 33 months
Population: Intent-To-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
Number analyzed (Participants) | 136 | 136
Months | 20.6 [14.4 to NA] — Not estimable due to insufficient number of participants with events | 19.4 [15.4 to 23.1]
Statistical Analysis 1: Comparison: Arm A (O+T+C) vs Arm B (P+T+C); Test type: Other; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.67 to 1.34] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: The number of participants who experienced TEAEs and SAEs was reported. An adverse event refers to any unintended or unfavorable sign, symptom, or condition (including abnormal lab results) that occurs during the study, regardless of whether it is linked to the study drug. Investigators evaluated the severity of each adverse event according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.
Time Frame: From first dose of study drug to 30 days after last dose, up to the study completion date cut-off date of 04 September 2024 (up to 32.4 months)
Population: The Safety Analysis Set included all randomized participants who received at least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
Number analyzed (Participants) | 135 | 136
Participants
  Number of participants with any TEAEs | 134 | 135
  Number of participants with SAEs | 63 | 74

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization up to study completion date cut-off date of 04 September 2024, up to 33 months. AEs are reported from first dose of study drug to 30 days after last dose, up to study completion date of 04 September 2024, up to 32.4 months.
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events are based on all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Arm A (O+T+C) | Arm B (P+T+C)
All-Cause Mortality (participants affected / at risk) | 63/136 | 70/136
Serious Adverse Events (participants affected / at risk) | 63/135 | 74/136
Other Adverse Events (participants affected / at risk) | 132/135 | 132/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (O+T+C) (N=135) | Arm B (P+T+C) (N=136)
Anaemia (Blood and lymphatic system disorders) | 4 (6) | 5 (5)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (5)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 3 (4)
Immune-mediated pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (6) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 4 (5)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Focal peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Haematological infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10) | 13 (15)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (7) | 3 (3)
Platelet count decreased (Investigations) | 3 (5) | 5 (5)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 5 (6) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pseudocellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (O+T+C) (N=135) | Arm B (P+T+C) (N=136)
Anaemia (Blood and lymphatic system disorders) | 90 (175) | 81 (142)
Leukopenia (Blood and lymphatic system disorders) | 11 (42) | 13 (40)
Lymphopenia (Blood and lymphatic system disorders) | 3 (11) | 5 (20)
Neutropenia (Blood and lymphatic system disorders) | 12 (19) | 11 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (17) | 8 (22)
Supraventricular extrasystoles (Cardiac disorders) | 5 (5) | 4 (7)
Hyperthyroidism (Endocrine disorders) | 10 (12) | 8 (10)
Hypothyroidism (Endocrine disorders) | 21 (23) | 16 (18)
Lacrimation increased (Eye disorders) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 13 (14)
Constipation (Gastrointestinal disorders) | 45 (65) | 40 (56)
Diarrhoea (Gastrointestinal disorders) | 21 (27) | 25 (28)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (6) | 5 (5)
Nausea (Gastrointestinal disorders) | 38 (50) | 51 (98)
Stomatitis (Gastrointestinal disorders) | 14 (15) | 8 (8)
Vomiting (Gastrointestinal disorders) | 24 (36) | 30 (59)
Asthenia (General disorders) | 12 (19) | 18 (28)
Fatigue (General disorders) | 27 (40) | 24 (31)
Malaise (General disorders) | 3 (3) | 9 (9)
Oedema peripheral (General disorders) | 11 (13) | 19 (22)
Pyrexia (General disorders) | 18 (22) | 20 (30)
COVID-19 (Infections and infestations) | 20 (24) | 15 (24)
Pneumonia (Infections and infestations) | 12 (18) | 14 (14)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 9 (11)
Urinary tract infection (Infections and infestations) | 4 (4) | 5 (6)
Alanine aminotransferase increased (Investigations) | 41 (69) | 43 (67)
Aspartate aminotransferase increased (Investigations) | 40 (75) | 37 (57)
Bilirubin conjugated increased (Investigations) | 4 (5) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 4 (6) | 6 (9)
Blood bilirubin increased (Investigations) | 8 (17) | 14 (15)
Blood creatine phosphokinase increased (Investigations) | 3 (4) | 6 (6)
Blood creatinine increased (Investigations) | 10 (10) | 22 (25)
Blood lactate dehydrogenase increased (Investigations) | 11 (19) | 8 (10)
Blood urea increased (Investigations) | 3 (4) | 5 (5)
Fibrin D dimer increased (Investigations) | 5 (6) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 5 (8) | 13 (17)
Lymphocyte count decreased (Investigations) | 22 (52) | 12 (47)
Neutrophil count decreased (Investigations) | 59 (188) | 50 (175)
Neutrophil count increased (Investigations) | 4 (6) | 5 (7)
Platelet count decreased (Investigations) | 51 (107) | 37 (64)
SARS-CoV-2 test positive (Investigations) | 13 (15) | 16 (17)
Weight decreased (Investigations) | 16 (20) | 18 (18)
Weight increased (Investigations) | 18 (23) | 14 (17)
White blood cell count decreased (Investigations) | 61 (196) | 54 (166)
Decreased appetite (Metabolism and nutrition disorders) | 37 (42) | 42 (55)
Dehydration (Metabolism and nutrition disorders) | 4 (25) | 6 (40)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5 (8) | 1 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (28) | 16 (19)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 (21) | 5 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (4) | 8 (18)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 30 (53) | 23 (34)
Hypocalcaemia (Metabolism and nutrition disorders) | 7 (10) | 6 (9)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (36) | 17 (24)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (11) | 6 (8)
Hyponatraemia (Metabolism and nutrition disorders) | 20 (36) | 21 (26)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 10 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (18) | 9 (10)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6)
Dizziness (Nervous system disorders) | 12 (16) | 7 (7)
Dysgeusia (Nervous system disorders) | 7 (7) | 4 (5)
Headache (Nervous system disorders) | 12 (16) | 12 (13)
Hypoaesthesia (Nervous system disorders) | 7 (7) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 12 (13)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (5)
Insomnia (Psychiatric disorders) | 16 (17) | 13 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (32) | 21 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 12 (13)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 8 (17) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 8 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 25 (25) | 26 (28)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (44) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 42 (62) | 27 (43)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Hypertension (Vascular disorders) | 4 (4) | 5 (5)
Hypotension (Vascular disorders) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT05014815/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/15/NCT05014815/SAP_001.pdf